CLINICAL TRIAL: NCT01141257
Title: A Phase I, Open-label Study of the Safety, Tolerability, and Pharmacokinetics of Angiocal® (PRS-050-PEG40) in Patients With Solid Tumors
Brief Title: Study of Angiocal® in Patients With Solid Tumors, Investigating Safety, Tolerability, Blood Concentration of Study Drug
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Pieris Pharmaceuticals GmbH (Industry)
Collaborators: FGK Clinical Research GmbH (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Pieris001
Record Dates: First submitted 2010-05-28; First posted 2010-06-10 (Estimated); Last update posted 2011-10-19 (Estimated); Status verified 2011-10

CONDITIONS: Solid Tumor
Keywords: Angiocal®; PRS-050-PEG40; Solid tumor; Phase I

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Angiocal® (Experimental): Angiocal®
  Interventions: Drug: Angiocal® (PRS-050-PEG40)

INTERVENTIONS:
Drug: Angiocal® (PRS-050-PEG40) — Single dose of Angiocal® i.v. (intravenous) on Day 1 and further applications of Angiocal® i.v. during a repeated dosing period.

SUMMARY:
The purpose of this study is to determine if Angiocal® (PRS-050-PEG40) is safe and well tolerated when it is injected into the veins of patients with solid tumors. Other purposes of this study are to investigate how the body of the patients reacts to Angiocal®, how the blood level of Angiocal® develops after injection and how the tumor responds to the injection of Angiocal®.

DETAILED DESCRIPTION:
This is a phase I, open-label, dose escalation study with Angiocal® in patients with solid tumors using a group sequential adaptive treatment assignment. Patients will be allocated to different dose levels in small cohorts and will receive one single dose application on Day 1, followed by a repeated dosing period. The primary objective of the study is to evaluate the safety and tolerability of Angiocal® when administered intravenously to patients with solid tumors. The secondary objectives of the study are the characterization of the pharmacodynamic response, evaluation of the pharmacokinetic profile of Angiocal®, observation of tumor response.

ELIGIBILITY:
Inclusion Criteria:

* Males or females with advanced, recurrent or metastatic cancer, refractory to standard therapy;
* Age ≥18 years;
* Signed informed consent form and ability to understand the study procedures.

Exclusion Criteria:

* Concomitant anticancer therapy, including radiation;
* Current or previous (within 30 days of first study dosing) treatment with another investigational drug or participation in another clinical study;
* Chronic daily treatment with aspirin (>325 mg/day) or clopidogrel (>75 mg/day);
* Chronic daily treatment with corticosteroids, with the exception of inhaled steroids;
* Inadequate bone marrow function;
* Inadequate liver function;
* Inadequate renal function;
* Patients not receiving anticoagulant medication who have an International Normalized Ratio (INR) >1.5 or an activated partial thromboplastin time (aPTT) >1.5 x ULN within 7 days prior to first study treatment;
* Patients with lymphomas;
* Evidence of spinal cord compression or brain metastases;
* Other malignancy diagnosed within the previous 5 years;
* Pregnant or lactating females.;
* All patients who do not use a highly effective method of birth control;
* Major surgical procedure (including open biopsy) within 28 days prior to the first study treatment, or anticipation of the need for major surgery during the course of the study treatment;
* Minor surgical procedures, within 24 hours prior to the first study treatment;
* History or evidence of inherited bleeding diathesis or coagulopathy with the risk of bleeding;
* Uncontrolled hypertension or clinically significant (i.e. active) cardiovascular disease;
* History of abdominal fistula, grade 4 bowel obstruction or gastrointestinal perforation, intra-abdominal abscess within 6 months of enrollment;
* Lung carcinoma of squamous cell histology or any histology in close proximity to a major vessel;
* Serious non-healing wound, peptic ulcer or bone fracture;
* Known hypersensitivity to the study medication or any of its excipients;
* Evidence of any other medical conditions that may interfere with the planned treatment, affect patient compliance or place the patient at high risk of treatment-related complications;
* Previous enrollment in this study;
* Known hepatitis B or C or HIV infection;
* Employees of the sponsor or patients who are employees or relatives of the investigator.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2010-05; Primary Completion 2011-09 (Actual); Study Completion 2011-09 (Actual)

PRIMARY OUTCOMES:
Dose limiting toxicity | Throughout the course of the study
  Dose limiting toxicity is determined by recording and evaluating adverse events / toxicity.

SECONDARY OUTCOMES:
Pharmacokinetic analysis | Throughout the course of the study
  AUC_0- τ; AUC_0-tlast; AUC_0-∞; C_max; T_max; t_½; CL; V_z; V_ss; RA_AUC; RA_Cmax; RL; dose normalized values (norm) for AUC_0-τ and C_max will be determined by dividing the original toxicokinetic parameter by the dose level.
Development of biomarkers in blood over time | Throughout the course of the study
Response of target lesions over time | Throughout the course of the study
  The objective tumor response for target lesions will be presented over time, employing the categories 'complete response', 'partial response, 'progressive disease´ and 'stable disease' and absolute changes.
ECOG performance status | Throughout the course of the study
  ECOG = Eastern Cooperative Oncology Group
Clinical laboratory measures | Throughout the course of the study
  Hematology, biochemistry, coagulation parameters, and urinalysis.
Anti-drug antibodies | Throughout the course of the study
Results of 12-lead Electrocardiogram by time point | Throughout the course of the study
  Changes from the baseline visit will be presented using shift tables (employing the categories 'normal', 'abnormal, clinically not significant' and 'abnormal, clinically significant') and absolute changes in laboratory values, if appropriate. Changes from the baseline visit in QTc between >30 and <60 ms and >60 ms will be listed and summarized separately.
Changes of vital signs from the baseline visit | Throughout the course of the study
  Heart rate, blood pressure and body temperature.
Physical examination | Throughout the course of the study
  Any changes in physical examination findings from baseline visit will just be summarized, since the physical examiniations will not result in measurable values.

CONTACTS AND LOCATIONS:
Overall Officials: Laurent Audoly, PhD, Study Director — Pieris Pharmaceuticals GmbH
Locations (2):
- Germany (2):
  - Breisgau, Baden-Wurttemberg
  - Ruhrgebiet, North Rhine-Westphalia

REFERENCES:
- [Derived] Mross K, Richly H, Fischer R, Scharr D, Buchert M, Stern A, Gille H, Audoly LP, Scheulen ME. First-in-human phase I study of PRS-050 (Angiocal), an Anticalin targeting and antagonizing VEGF-A, in patients with advanced solid tumors. PLoS One. 2013 Dec 13;8(12):e83232. doi: 10.1371/journal.pone.0083232. eCollection 2013. PMID 24349470